CLINICAL TRIAL: NCT02826928
Title: Diagnostic Performances of Urine and Plasma 5-hydroxyindolacetic Acid (5HIAA) Values in Patients With Small-intestine Neuroendocrine Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PO15138*
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2022-06

CONDITIONS: Small-intestine Neuroendocrine Tumors (Carcinoid Tumors)
MeSH Terms: conditions — Carcinoid Tumor

ARMS (2):
- patients with small-intestine neuroendocrine tumors (Experimental)
  Interventions: Biological: blood sample withdrawn
- control subjects with irritable bowel syndrome (Experimental)
  Interventions: Biological: blood sample withdrawn

INTERVENTIONS:
Biological: blood sample withdrawn

SUMMARY:
Urinary measure of 5-hydroxyindolacetic acid (5HIAA) is an important marker for the diagnosis and follow-up of patients with small-intestine neuroendocrine tumors. Although this marker has good specificity, its sensitivity is moderate and its dosage is constraining, since it requires urine collection over 2-3 days and specific diet. Preliminary data suggested that overnight 5HIAA value may be representative of 24-hour 5HIAA value, and that plasma 5HIAA dosage could be a valuable alternative to urine 5HIAA dosage. The main objective of this study is to compare sensitivity and specificity of overnight 5HIAA value, 24-hour 5HIAA value and plasma 5HIAA value, in patients with small-intestine neuroendocrine tumors.

DETAILED DESCRIPTION:
This study primarily aims at comparing the sensitivity and specificity of overnight 5HIAA value, 24-hour 5HIAA value and plasma 5HIAA value, in patients with small-intestine neuroendocrine tumors. Secondary objectives include the correlation of 5HIAA values with chromogranin A, carcinoid syndrome and tumor burden and the evaluation of the compliance to the diet and its correlation with 5HIAA values.

The study group will include patients with proven neuroendocrine tumors of various stages and functioning syndrome profile. A control group will be constituted with subjects having irritable bowel syndrome, in which a neuroendocrine tumor is ruled out. After providing informed consent, patients fitting with inclusion criteria will be included in the study. Patients will have to follow a specific diet, and interrupt/avoid certain medication, during the 2 days before and the 2 days during the sampling period. Whole urine samples will be collected during 2 consecutive days, in 4 parts (day1, night 1, day 2, night 2). Blood samples will be collected at the morning of days 2 and 3. Observance with diet and drug restriction will be evaluated at the morning of day 3.

ELIGIBILITY:
Inclusion criteria:

* Histologically proven small-intestine neuroendocrine tumors, at initial diagnosis or during the follow-up
* Irritable bowel syndrome, diagnosed following Rome III criteria, who had an ileo-colonoscopy and an abdominal CT-scan within the 12 last months
* Age > 18 years
* No antitumor treatment within the last three months excepted somatostatin analogs
* Ability of understanding and approving the study protocol and of providing written consent
* Affiliation to the French Health Social System

Exclusion criteria

* Small-intestine neuroendocrine tumor in remission (no detectable disease)
* Other malignancies than small-intestine neuroendocrine tumors (excepted if in remission for more than 2 years)
* Kidney insufficiency (MDRD < 60/min)
* Urinary incontinency or inability to collect urines
* Any antitumor treatment within the last three months excepted somatostatin analogs
* Inability to interrupt treatments interfering with 5HIAA dosage
* Pregnancy
* Patients under law protection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
urine 5HIAA value | 24-hour

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Result] de Mestier L, Savagner F, Brixi H, Do Cao C, Dominguez-Tinajero S, Roquin G, Goichot B, Hentic O, Dubreuil O, Hautefeuille V, Walter T, Cadiot G. Plasmatic and Urinary 5-Hydroxyindolacetic Acid Measurements in Patients With Midgut Neuroendocrine Tumors: A GTE Study. J Clin Endocrinol Metab. 2021 Mar 25;106(4):e1673-e1682. doi: 10.1210/clinem/dgaa924. PMID 33382891